CLINICAL TRIAL: NCT00146510
Title: HealtheLifestyle Behavioral Intervention Clinical Trial
Brief Title: HealtheTech Lifestyle Program
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Cooper Institute (Other)
Collaborators: HealtheTech (Unknown)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: CI-0126
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Obesity
Keywords: weight control; compliance; physical activity; nutrition; Health Behavior; Patient Compliance
MeSH Terms: conditions — Obesity; Patient Compliance; Motor Activity; Health Behavior

INTERVENTIONS:
Behavioral: HealtheLifestyle Program
Behavioral: step counters with monthly feedback on logs

SUMMARY:
The purpose of the study is to determine the efficacy of resting metabolic rate (RMR) using BodyGem and BalanceLog in helping overweight and obese individuals manage their weight.

DETAILED DESCRIPTION:
The study plans are to develop and test the efficacy of a practical, structured, and time-limited behavioral intervention (HealtheLifestyle Program) as a supplement to standard HealtheTech products. Approximately 130 participants will be recruited and randomized to either the HealtheTech Program (focusing on calorie and exercise goals using the BalanceLog for tracking), the HealtheLifestyle Program (using step counters, monthly email letters and calls providing information on activity, nutrition, and weight loss), or a delayed treatment program (after 3 months undergo the intervention above).

ELIGIBILITY:
Inclusion Criteria: healthy adult men and women, 18-60 years -

Exclusion Criteria: not currently participating in a structured diet or exercise program

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130
Dates: Start 2004-03; Study Completion 2006-02

PRIMARY OUTCOMES:
HealtheLifestyle participants will have greater weight loss

SECONDARY OUTCOMES:
HealtheLifestyle Program will increase efficacy of products

CONTACTS AND LOCATIONS:
Overall Officials: Heather Kitzman, MPH, Study Director — The Cooper Institute
Locations (1):
- The Cooper Institute, Dallas, Texas, United States